CLINICAL TRIAL: NCT05017779
Title: A Hybrid Effectiveness-implementation Trial of a School Based Executive Function Treatment for Transition Age Autistic Youth
Brief Title: A Hybrid Effectiveness-implementation Trial of a High School-based Executive Function Treatment for Autistic Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Lauren Kenworthy, Chief of Neuropsychology, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH124772 (NIH)
Record Dates: First submitted 2021-07-27; First posted 2021-08-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Executive Dysfunction; Autism Spectrum Disorder; Adolescent Behavior
Keywords: Autism Spectrum Disorder; Executive Functioning; Intervention; High school
MeSH Terms: conditions — Autism Spectrum Disorder; Adolescent Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Unstuck & On Target: High School) (Experimental): School staff will receive training on the Unstuck and On Target: High School (UOT:HS) curriculum, and deliver lessons to students during the school day. Interventionists will have the option to participate in ongoing check-ins with study staff. Parents are provided home extensions for each lesson and have the option to participate in trainings delivered by study staff to support generalization of skills to the home environment.
  Interventions: Behavioral: Unstuck & On Target: High School
- Usual Care (Other): Participants in schools assigned to the TAU condition will continue to receive the standard school-based Individualized Education Plan (IEP) accommodations and school supports that would typically be provided.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Unstuck & On Target: High School — Unstuck & On Target: High School (UOT:HS) is a group-based curriculum for high school students that targets executive function skills using Cognitive Behavior Therapy (CBT) techniques. UOT:HS focuses on key functions needed for adult success, such as: self-advocacy, flexibility, time management, motivation, goal setting, developing plans, monitoring progress. Guided practice begins with concrete interventionist support and moves to interventionist cueing, self-cueing, and finally automatic use of the skills without support. Lessons are delivered by school personnel within the school setting. Home extension activities are provided to parents.
  Other Names: Formerly Flexible Futures
  Arms: Intervention (Unstuck & On Target: High School)
Other: Treatment as Usual — Participants in schools assigned to the Treatment as Usual (TAU) condition will continue to receive the standard school-based IEP accommodations and school supports that would typically be provided. Data will be collected on the types of supports TAU schools offer, and what supports TAU students receive.
  Arms: Usual Care

SUMMARY:
This study will test the effectiveness of a school-based cognitive behavioral executive function (EF) intervention, Unstuck & On Target High School (UOT:HS), for transition-age youth with autism spectrum disorder (ASD). UOT:HS was designed to be embedded in high schools and delivered by school staff to improve generalization of skills, increase access to mental health care, and fill a gap in evidence-based approaches to support postsecondary transition. UOT:HS targets flexibility and planning skills and focuses on key functions needed for adult success across 25, 1-hour lessons. School staff will be trained to deliver UOT:HS, study staff will provide ongoing check-ins, and parents will be offered home extensions for each lesson and two trainings to generalize skills to the home environment. Behavioral and parent-report data will be collected prior to intervention, post-intervention, and at 4-to-6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive/Behavioral capacity to benefit and understand Unstuck material as determined by teacher guided by probes related to pragmatic language that align with verbal demands of the curriculum.
2. Evidence of autism supported by at least one of the following:

   * Eligible and/or receiving school-based services or supports for autism
   * Prior clinical diagnosis of autism from a qualified health professional (as indicated by parent report)
   * Demonstrates characteristics of autism consistent with DSM-5, as judged by a clinical autism expert, based on all available information gathered through the screening, consenting, and testing process (including information gathered through the Social Communication Questionnaire via parent/teacher report, and SRS-2,)
3. Capacity to benefit and understand unstuck material as determined by teacher

Exclusion Criteria:

1. Students must have a level of proficiency in English to complete questionnaires and study procedures in English. Parents must have a level of proficiency in English or Spanish to complete questionnaires and study procedures in English or Spanish.
2. Student is not able to participate in UOT:HS due to their schedule or ability to benefit from curriculum material as determined by teacher.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Classroom Behavior | Baseline to End of Intervention (up to end of academic year, approx 9 months)
  Change in Classroom Behavior will serve as the primary outcome at end of intervention. Classroom behavior will be assessed through 15-minute classroom observations conducted by a trained research staff member masked to treatment condition. Observations will occur during the school day in an academic (non-intervention) class. Raters use a standardized form to detect the presence or absence of seven observable behaviors: social appropriateness, on task behavior, initiation, transitions, organization, getting stuck/preservation, expression of overwhelm/negativity.
Adaptive Behavior (at follow-up) | Baseline, End of Intervention, Follow-up (approx. 6 months after end of intervention)
  Change in adaptive behavior will serve as the primary outcome at follow-up (e.g., approximately six month after end of intervention). Adaptive behavior will be measured via parent-report on the Adaptive Behavior Assessment System, Third Edition (ABAS-3). The ABAS-3 is a well-validated parent report measure that assesses practical, everyday skills needed to effectively and independently take care of oneself and interact with others across the lifespan. Performance is represented as standard scores, with higher scores indicating better adaptive skills.

SECONDARY OUTCOMES:
Adaptive Behavior (end of intervention) | Baseline, End of Intervention (up to end of academic year, approx 9 months)
  Change in adaptive behavior will serve as the secondary outcome at the end of intervention. Adaptive behavior will be measured via parent-report on the Adaptive Behavior Assessment System, Third Edition (ABAS-3). The ABAS-3 is a well-validated parent report measure that assesses practical, everyday skills needed to effectively and independently take care of oneself and interact with others across the lifespan. Performance is represented as standard scores (mean=100; SD=15), with higher scores indicating better adaptive skills.

OTHER OUTCOMES:
Executive Function Challenge Task (EFCT) | Baseline to End of Intervention (up to end of academic year, approx 9 months)
  The "Executive Function Challenge Task" (EFCT) is an objective and ecologically valid task developed by our research team to assess flexibility and planning skills in a social context conducted by a trained research staff member masked to treatment condition. The EFCT uses a standardized, semi-structured protocol which does not provide explicit rules for completing the tasks to mimic the implicit, unspoken, unstructured expectations in everyday life. The EFCT consists of challenges across several activities and responses are scored on a 3-point scale for each task. The scale (0-good, 1-intermediate, 2-poor performance) has task-specific behavioral markers to guide scoring.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | Baseline, End of Intervention, Follow-up (approx. 6 months after end of intervention)
  The "Behavior Rating Inventory of Executive Function, Second Edition" (BRIEF-2) is a well-established parent-report measure of real-world EF skills, with the Shift subscale measuring cognitive flexibility.
Dimensional Change Card Sort - NIH Toolbox | Baseline to End of Intervention (up to end of academic year, approx 9 months)
  The Dimensional Change Card Sort (DCCS) (NIH Toolbox) is a 4-minute, standard lab-based task for assessing cognitive flexibility in terms of set-shifting. Participants are required to sort a series of bivalent cards first according to one dimension (e.g., color) and then according to another (e.g., shape). It is normed from ages 4-85.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Kenworthy, PhD, Principal Investigator — Children's Research Institute, Children's National Hospital
Locations (1):
- Center for Autism Spectrum Disorders, Children's National Hospital, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared via the National Institute of Mental Health's National Data Archive (NDA).
Time Frame: Descriptive/raw de-identified data will be reported semi-annually through NDA.
Access Criteria: Request login access to NDA data